CLINICAL TRIAL: NCT06952491
Title: Research and Engagement on Substance Use: Harnessing Awareness and Personalized Education (RESHAPE) to Improve Well-being and Self-efficacy
Acronym: RESHAPE
Status: Enrolling by invitation | Type: Observational
Sponsor: Evidation Health (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00085294; 1R44DA062284-01 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Substance Use Disorder (SUD)
Keywords: Substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with self-reported substance use disorder or at risk for substance use disorder: Participants from the Evidation platform with self-reported substance use disorder or at risk for substance use disorder as defined by cannabis use, tobacco use, illegal drug use, or prescription medication use for nonmedical reasons on at least 2-3 times in the past year Self-reports at least one of the following health-related social needs as assessed by American Academy of Family Physicians Social Needs Screening Tool
  * Housing instability
  * Non-reliable transportation
  * Food insecurity
  * Utility needs
  * Personal safety

SUMMARY:
The goal of this study is to gather feedback on a potential program that collects and shares real-world information to help create products and services to support people who have substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* U.S. resident
* Speaks, read, and understands English
* Adults ≥ 21 years of age
* Self-reported substance use disorder or at risk for substance use disorder as defined by cannabis use, tobacco use, illegal drug use, or prescription medication use for nonmedical reasons on at least 2-3 times in the past year
* Self-reports at least one of the following health-related social needs as assessed by American Academy of Family Physicians Social Needs

Screening Tool:

* Housing instability
* Non-reliable transportation
* Food insecurity
* Utility needs
* Personal safety
* Willingness and availability to participate in a recorded online interview (Phase 1A participants)

Exclusion Criteria:

* Participation in Phase 1A (among Phase 1B participants), to be assessed using participation history

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: United States residents
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Willingness to participate in a future substance use disorder program | Baseline
  Number and percentage of interview and survey respondents reporting willingness to participate in a future substance use disorder program
Perceived usefulness and expected use of a future program's potential features and content | Baseline
  Number and percentage of interview and survey respondents reporting that the future program's potential features are useful
To quantify and describe real-world health related social needs and/or substance use and/or demographics survey(s) previously collected on the Evidation platform | From approximately 1 year prior to enrollment until study enrollment
  Number and percentage of interview and survey respondents who completed at least one health related social needs and/or substance use and/or demographics survey on the Evidation platform in the past year
Perceived expected use of potential features and content to be included in a program to improve well-being and self-efficacy for health promoting activities | Baseline
  Number and percentage of interview and survey respondents reporting that they expect to use each of the future program's potential features and content
To quantify and describe real-world data from a connected wearable device previously collected on the Evidation platform | From approximately 1 year prior to enrollment until study enrollment
  Average number of days with valid steps, sleep, and heart rate data from a connected wearable device in the past year
To quantify and describe real-world data from responses to daily mood, stress, and sleep diaries previously collected on the Evidation platform | From approximately 1 year prior to enrollment until study enrollment
  Average number of days with responses to daily mood, stress, and sleep diaries in the past year

CONTACTS AND LOCATIONS:
Overall Officials: Christian Cerrada, PhD, Principal Investigator — Evidation Health
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Taylor B, Henshall C, Kenyon S, Litchfield I, Greenfield S. Can rapid approaches to qualitative analysis deliver timely, valid findings to clinical leaders? A mixed methods study comparing rapid and thematic analysis. BMJ Open. 2018 Oct 8;8(10):e019993. doi: 10.1136/bmjopen-2017-019993. PMID 30297341
- [Background] Schuler MS, Prince DM, Collins RL. Disparities in Social and Economic Determinants of Health by Sexual Identity, Gender, and Age: Results from the 2015-2018 National Survey on Drug Use and Health. LGBT Health. 2021 Jul;8(5):330-339. doi: 10.1089/lgbt.2020.0390. Epub 2021 Jun 8. PMID 34101498